Title: Intelligent Personal Assistant for Managing Depression in Homebound Older Adults

NCT Number: NCT04900272

Document Date: February 25, 2022

## **Verbal Consent to Participate in Research**

**Title of Research Study:** Intelligent Personal Assistant for Managing Depression in Homebound Older Adults

IRB Study Number: STU00212384

Principal Investigator: Katherine O'Brien, MD

**Supported By:** This research is supported by the Claude D. Pepper Older Americans Independence Center at Northwestern University and the National Institute on Aging.

**Introduction:** I am \_\_\_\_\_\_, a doctoral student in the Department of Psychiatry at Northwestern University.

#### **Key Information about this research study:**

The following is a short summary of this study to help you decide whether to be a part of this study. The purpose of this study is to design a companion booklet and pilot test it with voice-controlled intelligent personal assistants (VIPA), like Google Home or Amazon Alexa, to provide homebound older adult patients with skills and tools to help manage social isolation. Homebound is defined as a person who is unable to leave the home without assistance of a device (such as a walker, wheelchair or cane) or another person, due to any physical or cognitive condition. The companion booklet is a document that will be created using feedback obtained from a panel of geriatric experts, highlighting features of the VIPA that may be most beneficial to socially-isolated older adults.

You will be asked to utilize a Google Home or Amazon Alexa VIPA device and companion booklet for 16 weeks in order to identify whether a Google Home or Amazon Alexa device may a useful tool for homebound older adults who may be socially isolated. At the beginning of the study, someone from our research team will visit your home to set up the device and review the companion booklet with you, or someone will assist you virtually with the set up. Then, during the 16 week period, you will be surveyed over the phone, online, or in-person four times to complete various surveys about aspects of your health and well-being, as well as. You will also be asked to provide feedback on your experience with the device and booklet.

We expect that you will be in this research study for approximately 6 months although you will not be engaged in the study during that entire time. You will use the Google Home or Amazon Alexa VIPA device and companion booklet for a 16 week period. You will be asked to complete four telephone, online, or in-person surveys, which will take place at the beginning of the period, after 4 weeks, after 8 weeks, and after 16 weeks. These surveys will ask you about your experience using the device and booklet, as well as questions about your health and well-being.

The primary risk of participation is that using a VIPA may result in a loss of confidentiality if someone else were to access the information gathered by the Google Home or Amazon Alexa device. Additionally, you may feel uncomfortable answering some questions related to your health and wellbeing. If this does happen or any questions make you feel uncomfortable and you prefer not to answer, you may skip them.

The main benefit of participation is that you may gain a better understanding of how to use a voice-controlled personal assistant.

Version date: August 26, 2021 HRP-1709 / v05132019

## **Verbal Consent to Participate in Research**

#### Here is why you are being asked to take part in this research study:

I am asking you to take part in this research study because you are an adult aged 65 years or older who is a homebound patient and is English-speaking.

#### This is what you should know about being in a research study

- Whether or not you take part is up to you.
- You can choose not to take part. You can also agree to take part and later change your mind.
- Your decision will not be held against you.
- You can ask all the questions you want before you decide.

### If you say that "Yes, you want to be in this research," here is what you will do

During the study, we will ask you to use the Google Home or Amazon Alexa device and its companion booklet over a 16 week period. During this period, you will be asked to complete four telephone, online, or in-person surveys, which will take place at the beginning of the period, after 4 weeks, after 8 weeks, and after 16 weeks. These surveys will ask you about your experience using the device and booklet, as well as questions about your health and well-being.

#### If you say that you do not want to be in this research:

You can decide not to participate in this research and it will not be held against you.

### You can say "Yes," but change your mind later

You can leave the research at any time and it will not be held against you. We can end the interview at any time. Just let me know if you want to do this. If this happens, I will ask you if any data collected up until that point may be used in the research.

# This is what will happen to the information collected for this research

Efforts will be made to limit the use and disclosure of your personal information, including research study records, to people who have a need to review this information. We cannot promise complete secrecy. Organizations that may inspect and copy your information include the IRB and other representatives of this institution.

## Here is some other information that is useful for you to know

If you agree to take part in this research study, we will provide you with the Google Home VIPA device which you will use during the course of the study. As a thank you for your time, you will keep the device after your participation in the study is complete (estimated value of \$40). You will also receive a \$20 gift card at the end of the study. You will receive the gift card compensation by mail.

## Here is who you can talk to

If you have questions, concerns, or complaints talk to the Principal Investigator, Dr. Katie O'Brien at katherine.obrien@northwestern.edu. This research has been reviewed and approved by an Institutional Review Board ("IRB"). You may talk to them at (312) 503-9338 or <a href="mailto:irb@northwestern.edu">irb@northwestern.edu</a> if:

- Your questions, concerns, or complaints are not being answered by the research team.
- You cannot reach the research team.
- You want to talk to someone besides the research team.

Version date: August 26, 2021 HRP-1709 / v05132019

IRB #: STU00212384 Approved by NU IRB for use on or after 2/25/2022 through 2/24/2023.

## **Verbal Consent to Participate in Research**

- You have questions about your rights as a research participant.
- You want to get information or provide input about this research.

## **Optional Elements:**

The following research activity is optional, meaning that you do not have to agree to it in order to participate in the research study. Please indicate your willingness to participate in this optional activity by saying "Agree" or "Disagree".

The researcher may contact me in the future to see whether I am interested in participating in other

| research studies by the investigator | r of this study | 7. |
|---|---|---|
| Record participant's response: | Agree | Disagree |
| Consent: | | |
| | participant re | cord participant's response: _[NOTE: If a person esponse and the person's name is documented in your n.] |
| If response is Yes, then enter the P | articipant Na | me below |
| Participant Name (Printed) | | |
| Signature of person obtaining cons | sent | Date |
| Printed name of person obtaining of | consent | |
| 1 0 | | |

Version date: August 26, 2021 HRP-1709 / v05132019 IRB #: STU00212384 Approved by NU IRB for use on or after 2/25/2022 through 2/24/2023.

# Verbal Consent to Participate in Research

Version date: August 26, 2021 HRP-1709 / v05132019